CLINICAL TRIAL: NCT04315883
Title: Clinical Outcomes and Quality of Life After Transarterial Radioembolization With Yttrium-90 (TARE-Y90) in Children, Adolescents, and Young Adults With Liver Tumors
Brief Title: Yttrium-90 (TARE-Y90) in Children, Adolescents, and Young Adults With Liver Tumors
Status: Terminated | Type: Observational
Why Stopped: PI left organization and discontinued study
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: NEMOURS TARE-Y90: ST1901
Record Dates: First submitted 2020-03-02; First posted 2020-03-20 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Hepatoblastoma; Hepatocellular Carcinoma; Rhabdoid Tumor of Liver; Undifferentiated (Embryonal) Sarcoma of the Liver; Pediatric Liver Cancer; Liver Tumors
Keywords: Hepatoblastoma; Hepatocellular carcinoma; Rhabdoid tumor of the liver; Undifferentiated sarcoma of the liver; Liver transplant; unresectable; yttrium 90; Y90; radioembolization; resection; pediatric; cancer; liver tumor
MeSH Terms: conditions — Hepatoblastoma; Carcinoma, Hepatocellular; Disorders of Sex Development; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard Treatment: Evaluation of change of HRQOL survey responses will be performed:
  * at baseline (time of treatment) and
  * 1 month post treatment
  * 6 months post treatment
  * 12 months post treatment
  * 5 years post-treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
  Interventions: Behavioral: Quality of Life Assessment; Radiation: Transarterial Radioembolization

INTERVENTIONS:
Behavioral: Quality of Life Assessment — Evaluation of change of HRQOL survey responses will be performed:
  * at baseline (time of treatment) and
  * 1 month post treatment
  * 6 months post treatment
  * 12 months post treatment
  * 5 years post-treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Radiation: Transarterial Radioembolization — Deliver catheter directed yttrium-90 directly to liver tumors and assess -Progression Free Survival - Local and Metastatic
  * Local Tumor Response by calculating the decreases in tumor size and enhancement after treatment. This will be assessed by modified Response Evaluation Criteria for Solid Tumors (mRECIST).
  * Resection Rate following treatment
  * Transplant Rate following treatment
  * Histologic Response by assessing tumor histopathology in patients who undergo tumor resection or liver transplant
  * Biologic Response by monitoring serum tumor markers (e.g. alphafetoprotein-AFP) in AFP secreting tumors
  * Review of clinical course post-treatment-rehospitalization rate

SUMMARY:
This study will be performed to evaluate the Clinical Outcomes and Quality of Life after Transarterial Radioembolization with Yttrium-90 (TARE-Y90) in Children, Adolescents, and Young Adults with Liver Tumors. The treatment and techniques used here are well established in adults.

The purpose of this study is to evaluate:

1. the response to treatment and clinical outcomes of treatment with TARE Y-90 as part of standard therapy and
2. to assess the change in the patient's quality of life before, during and after treatment with TARE-Y90

DETAILED DESCRIPTION:
* Referral to Nemours Liver Tumor Program is made by the primary team (oncologist/surgeon).
* Phone discussion between the Nemours Liver Tumor Program Team will occur with the referring team about the patient.
* Phone call between the Nemours Liver Tumor Program Team and the family will occur prior to any visit to discuss the potential plan of care and the basics of the TARE-Y90 procedure and the Quality of Life surveys.

Review of medical records provided by referring institution will be done by the Nemours Liver Tumor Program Team including:

History, Scans-actual imaging required, Path report-slide submission required, Roadmaps, Labs, Other pertinent medical history and records

-Visit to Nemours/AI DuPont Children's Hospital for initial consultation will be arranged by the Nemours Liver Tumor Program Team.

The patient and family will meet with the team including:

Liver transplant surgeon (Dr Dunn), Interventional Radiologist (Dr Aguado), Social worker, Child life specialist, Pediatric oncologist (Dr Gresh - on site, Dr Katzenstein by telemedicine)

* Attempt will be made to schedule the pre-planning angiogram as part of initial visit (2nd day of visit). The angiogram requires the following 3-4 hours (mapping of blood vessels in and around tumor - determines whether patient can receive Y90, Angiogram is done with the patient sedated and having been after midnight the night before, The patient is expected to be discharged on the same day of the angiogram- no admit is planned but occasionally the patient may need overnight observation to occur due to age of the patient or the length of the procedure.
* Return to home.
* Potential additional single cycle of chemotherapy may be given prior to return to Nemours for Y90.

All further Chemotherapy Care is coordinated with Nemours Liver Tumor oncologists

-A 2nd visit to AIDHC will occur for TARE-Y90 treatment: The procedure lasts about 2-3 hours. There is no planned admit but possible if any problems occur.

* 2 weeks post procedure a phone call follow-up after treatment will occur with the Nemours team
* 2 weeks post procedure the patient may resume chemotherapy when cleared by the Nemours team
* 4-6 weeks post Y90 treatment - a repeat CT/MRI will be done as well as lab tests.
* If possible, the CT/MRI to be done at AIDHC/Nemours but can be done locally if travel barriers exist.
* If the tumor is now resectable, planning will be made for resection at AIDHC/Nemours.
* Evaluation and change of HRQOL survey responses will be performed at baseline (time of treatment) and 1, 6, 12 months and 5 years post-treatment. These surveys will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls age < 21 years of age
* History of liver tumor
* Meet criteria for treatment with TARE-Y90

Exclusion Criteria:

* • Inability to complete required study procedures.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and Young adult patients with liver tumors
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Determine the impact of TARE-Y90 treatment on health related quality of life (HRQOL) | Assessed at baseline/time of treatment
  Evaluation of change of HRQOL survey responses will be performed:
  -at baseline (time of treatment)
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Determine the impact of TARE-Y90 treatment on health related quality of life (HRQOL) | Assessed at 1 month post therapy
  Evaluation of change of HRQOL survey responses will be performed:
  - 1 month post treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Determine the impact of TARE-Y90 treatment on health related quality of life (HRQOL) | Assessed at 6 months post therapy
  Evaluation of change of HRQOL survey responses will be performed:
  - 6 months post treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Determine the impact of TARE-Y90 treatment on health related quality of life (HRQOL) | Assessed at 12 months post therapy
  Evaluation of change of HRQOL survey responses will be performed:
  - 12 months post treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Determine the impact of TARE-Y90 treatment on health related quality of life (HRQOL) | Assessed at 5 years post therapy
  Evaluation of change of HRQOL survey responses will be performed:
  - 5 years post-treatment
  The HRQOL will be done by phone, mail or email. Responses will be captured and entered into a REDCAP database
Evaluate the efficacy and clinical utility of TARE-Y90 by examining 2 year survival | Patients will be assessed at 2 years post therapy
  Deliver catheter directed yttrium-90 directly to liver tumors and assess -Progression Free Survival - Local and Metastatic
  -
Evaluate the efficacy and clinical utility of TARE-Y90 by examining 5 year survival | Patients will be assessed at 5 years post therapy
  Deliver catheter directed yttrium-90 directly to liver tumors and assess -Progression Free Survival - Local and Metastatic
Evaluate the efficacy and clinical utility of TARE-Y90 by examining local tumor response | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Local Tumor Response by calculating the decreases in tumor size and enhancement after treatment. This will be assessed by modified Response Evaluation Criteria for Solid Tumors (mRECIST).
Evaluate the efficacy and clinical utility of TARE-Y90 by examining resection rate | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment.
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Resection Rate following treatment
Evaluate the efficacy and clinical utility of TARE-Y90 by examining Transplant rate | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment.
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Transplant Rate following treatment
Evaluate the efficacy and clinical utility of TARE-Y90 by examining histologic response | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment.
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Histologic Response by assessing tumor histopathology in patients who undergo tumor resection or liver transplant
Evaluate the efficacy and clinical utility of TARE-Y90 by examining biologic response | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment.
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Biologic Response by monitoring serum tumor markers (e.g. alphafetoprotein-AFP) in AFP secreting tumors
Evaluate the efficacy and clinical utility of TARE-Y90 by examining clinical course | Patients will be assessed at the end of treatment which is typically 2-4 months following treatment.
  Deliver catheter directed yttrium-90 directly to liver tumors and assess
  -Review of clinical course post-treatment-rehospitalization rate

CONTACTS AND LOCATIONS:
Overall Officials: Howard Katzenstein, Principal Investigator — Nemours
Locations (2):
- United States (2):
  - Nemours-AI duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Specialty Care, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aguado A, Ristagno R, Towbin AJ, Gupta A, Haberle S, Qi Z, Patel MN, Kukreja KU, Tiao GM, Geller JI. Transarterial radioembolization with yttrium-90 of unresectable primary hepatic malignancy in children. Pediatr Blood Cancer. 2019 Jul;66(7):e27510. doi: 10.1002/pbc.27510. Epub 2018 Nov 8. PMID 30406959